CLINICAL TRIAL: NCT07032389
Title: Polypill Strategy for the Treatment of Patients After Acute Coronary Syndromes - A Multicenter Randomized Controlled Trial
Brief Title: A Polypill for Acute Coronary Syndrome
Acronym: PolyACS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0861
Record Dates: First submitted 2025-06-19; First posted 2025-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Polypill; Adherence
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: The patient will be randomized into one of two groups: the polypill arm, receiving a 3-in-1 capsule containing dual antiplatelet therapy (DAPT) and a statin; or the usual care arm, receiving standard DAPT and statins as separate medications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Polypill (Experimental): The polypill combines DAPT and a high intensity statin: (a) aspirin 81 mg, (b) rosuvastatin (40 or 10 mg) and (c) prasugrel 10 mg or clopidogrel 75 mg.
  Interventions: Combination Product: Polypill
- Usual care (No Intervention): Participants in the usual care arm will be prescribed DAPT and statins as standard therapy in individual pills.

INTERVENTIONS:
Combination Product: Polypill — The polypill is an inert capsule designed to combine multiple individual medications into a convenient, once-daily pill. In this case it will include DAPT and a statin.
  Arms: Polypill

SUMMARY:
The current study aims to investigate whether combining the standard medications prescribed after acute coronary syndrome (ACS)-aspirin, P2Y12 inhibitors, and statins-into a single polypill can improve outcomes following an ACS event. Although these therapies are effective, gaps in adherence and uptake significantly contribute to risk or adverse events in the post-ACS period. This study is designed as a pragmatic, multi-center, randomized trial to assess the feasibility and effectiveness of a polypill-based strategy for treatment of ACS.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) poses a major public health challenge in the United States. ACS, a constellation of acute cardiovascular conditions including ST-segment elevation myocardial infarction (STEMI), non-ST-segment elevation myocardial infarction (NSTEMI), and unstable angina, is a major determinant of morbidity and mortality across the United States. An American will suffer from an ACS event every 40 seconds, and ~1 million individuals have an ACS event annually. The absolute 30-day and 1-year mortality rates following an ACS event have remained high over the past several years. Myocardial infarction, a component of ACS, is one of the five most expensive admission diagnoses, with an estimated cost to the US health system of $12.1 billion annually.

The risk of major adverse cardiac events or death is high in the immediate post-ACS period. Despite effective pharmacotherapies and early revascularization, patients with ACS remain at an increased risk of post-MI complications, including recurrent ischemic events, heart failure, mechanical complications, and death in the first few weeks following the index event. The rate of major adverse cardiovascular events (MACE) is six-fold higher within the first 30 days compared with one-year post-discharge from the index MI event (41% vs. 6.4%, annualized).The 30-day risk-adjusted mortality following an ACS event in the U.S. is among the highest among developed countries, ranging from 12% (NSTEMI) to 18% (STEMI). These observations highlight the need for more aggressive implementation of evidence-based therapies in the post-ACS period.

Significant gaps exist in the optimal utilization of evidence-based therapies post-ACS. Treatment for ACS includes urgent revascularization followed by initiation of dual antiplatelet therapy (DAPT), which includes aspirin, a P2Y12 inhibitor, and a high-intensity statin. While rates of percutaneous coronary intervention (PCI) following an ACS event have increased substantially over the past two decades, utilization of evidence-based medical therapies, specifically DAPT and high-intensity statin therapy, in the post-MI period are suboptimal. Low utilization rates may reflect physician factors (such as inadequate prescribing) and/or patient factors (low adherence). Evidence from clinical registries suggests that low adherence may play the larger role, as the vast majority of post-ACS patients are prescribed DAPT and statins (>90% prescription rates). For example, in the TRANSLATE-ACS registry, a multicenter study of MI patients treated with PCI, approximately one-third of patients reported suboptimal adherence to prescribed cardiovascular medications in the first six weeks after their hospitalization. Similarly, in the multicenter ACTION Registry-GWTG (Acute Coronary Treatment and Intervention Outcomes Network Registry-Get with the Guidelines) cohort of ~20,000 patients with ACS, the rates of non-adherence to P2Y12 and statin therapy within 90 days of the index event, assessed by the proportion of days covered (PDC), was 28% and 37%, respectively. Furthermore, non-adherence rates increase over time, reaching up to 50% by 12 months following the index ACS event.

Premature discontinuation of evidence-based therapies following an ACS event markedly increases the risk of an adverse event. Discontinuation of cardiac medications is associated with an increased risk of in-stent thrombosis, recurrent MI, and death, making optimal adherence in the subacute phase after ACS critical. For instance, among patients with an ACS event treated with a drug-eluting stent, premature discontinuation of P2Y12 inhibitor therapy is associated with a 9-fold higher risk of death. In-stent thrombosis is a severe complication with up to 45% risk of mortality, and the highest risk is within 30 days after stent placement. Discontinuing statin therapy after MI is associated with a 3-fold higher risk of death over a 1-year follow-up period.

There are important disparities in ACS outcomes by race and socioeconomic status. While the overall incidence of MI has declined over time, racial/ethnic disparities have persisted, with a higher risk of adverse outcomes among ACS patients of self-reported Black or Hispanic race/ethnicity. Black and Hispanic patients who present with ACS are younger on average and more likely to be uninsured and have less education. The risk of 30-day and 1-year mortality following an ACS event is significantly higher among patients of self-reported Black or Hispanic race/ethnicity (vs. white). In addition to racial/ethnic disparities, significant disparities in ACS outcomes have also been reported based on socioeconomic status. Specifically, individuals with low (vs. high) income or education levels and those living in socioeconomically disadvantaged neighborhoods have a higher risk of adverse outcomes following an ACS event. These disparities are driven by poor access to care, lower rates of revascularization, and less use of evidence-based therapies following an ACS.

DAPT and high-intensity statin utilization rates following an ACS event are lowest in patients from under-represented minority groups. Prior studies have demonstrated up to 20% lower adherence to P2Y12 inhibitors among patients of Black and Hispanic race/ethnicity within the six months following an ACS event. In addition, financial hardship and low SES are associated with lower self-reported adherence to evidence-based therapies within six weeks of an ACS. These data highlight the need for novel approaches to improve adherence to evidence-based therapies following an ACS event among Black and Hispanic individuals and those with socioeconomic disadvantages.

Polypill-based strategies reduce the risk of major adverse cardiovascular events in the primary and secondary prevention setting. Low-dose, multi-drug combinations of cardiovascular therapies have been examined to prevent cardiovascular outcomes in multiple primary and secondary prevention trials, including HOPE-3, TIPS-3, the PolyIran study, and most recently, the SECURE trial. It has been proposed that the benefits of a polypill approach are attributable to better patient adherence and reduced physician inertia. In the SECURE trial, patients with recent MI who were treated with a polypill containing aspirin, ramipril, and atorvastatin had a ~25% lower risk of cardiovascular death, nonfatal MI, or urgent coronary revascularization. Further, improvements in medication adherence and treatment satisfaction were documented in the polypill group compared with usual care.

Our research group has previously shown that a polypill-based strategy is feasible in low-income populations. Our group completed the largest U.S. trial to date investigating a polypill approach for the primary prevention of heart disease. In this trial, individuals at a federally-qualified community health center were randomized to a polypill versus usual care. Individuals in the polypill group had significant reductions in systolic blood pressure (-7 mm Hg, 95% CI: -2 to -12; p=0.003) and LDL cholesterol (-11 mg/dl, 95% CI: -5 to -18; p=0.0003), compared with those randomized to usual care. Two-thirds of participants had an income < $15,000.

While prior studies have demonstrated the efficacy of a polypill-based strategy in primary and secondary prevention, the polypill has not been evaluated for managing patients in the post-ACS setting. Patients are particularly vulnerable in the subacute period immediately following an ACS hospitalization due to the risk of stent thrombosis or other ischemic events. Moreover, prior polypill trials in the secondary prevention setting have focused on anti-hypertensive drugs, aspirin, and statins. Thus, there is a critical implementation gap related to non-adherence to P2Y12 inhibitors, one of the most essential therapies for managing ACS patients in the post-PCI subacute phase.

Given the significant pill burden for post-ACS patients, a polypill approach for patients in the subacute period following PCI may have substantial advantages. Thus, will conduct a pragmatic, open-label, Type 1 hybrid efficacy-implementation, multicenter clinical trial of a polypill-based strategy in post-ACS patients. The polypill will consist of a high-intensity statin, aspirin 81 mg, and a P2Y12 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Hospitalization for acute coronary syndrome with percutaneous coronary intervention
* Discharged on aspirin, prasugrel or clopidogrel, and a high-intensity statin

Exclusion Criteria:

* Current need for systemic anticoagulation
* Contraindication to receive any components of the polypill
* History of allergic reaction or intolerance to aspirin, prasugrel or clopidogrel, or rosuvastatin
* Comorbidities that might be expected to limit lifespan within the 12-month study period
* Increased risk of bleeding or planned urgent surgery that would necessitate use of DAPT for < 12 months
* Inability to provide written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Win ratio | 12-months
  The win ratio will include all-cause death, in-stent thrombosis, ischemic events (MI, hospitalization for unstable angina, unplanned revascularization), and bleeding events (hospitalization or ED visit for bleeding, red blood cell transfusion, or a bleeding event that leads to cessation of DAPT)

SECONDARY OUTCOMES:
Medication adherence | 12-months
  Medication adherence will be evaluated with the Morisky Medication Adherence Score (MMAS) and pill counts
Treatment satisfaction | 12-months
  Treatment satisfaction will be measured using the validated Treatment Satisfaction Questionnaire for Medication (TSQM)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):e344-426. doi: 10.1161/CIR.0000000000000134. Epub 2014 Sep 23. No abstract available. PMID 25249585
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention, 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery, 2012 ACC/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease, 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction, 2014 AHA/ACC Guideline for the Management of Patients With Non-ST-Elevation Acute Coronary Syndromes, and 2014 ACC/AHA Guideline on Perioperative Cardiovascular Evaluation and Management of Patients Undergoing Noncardiac Surgery. Circulation. 2016 Sep 6;134(10):e123-55. doi: 10.1161/CIR.0000000000000404. Epub 2016 Mar 29. No abstract available. PMID 27026020
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Okkonen M, Havulinna AS, Ukkola O, Huikuri H, Pietila A, Koukkunen H, Lehto S, Mustonen J, Ketonen M, Airaksinen J, Kesaniemi YA, Salomaa V. Risk factors for major adverse cardiovascular events after the first acute coronary syndrome. Ann Med. 2021 Dec;53(1):817-823. doi: 10.1080/07853890.2021.1924395. PMID 34080496
- [Background] Islek D, Alonso A, Rosamond W, Kucharska-Newton A, Mok Y, Matsushita K, Koton S, Blaha MJ, Ali MK, Manatunga A, Vaccarino V. Differences in incident and recurrent myocardial infarction among White and Black individuals aged 35 to 84: Findings from the ARIC community surveillance study. Am Heart J. 2022 Nov;253:67-75. doi: 10.1016/j.ahj.2022.05.020. Epub 2022 Jun 1. PMID 35660476
- [Background] Bradley EH, Herrin J, Wang Y, McNamara RL, Webster TR, Magid DJ, Blaney M, Peterson ED, Canto JG, Pollack CV Jr, Krumholz HM. Racial and ethnic differences in time to acute reperfusion therapy for patients hospitalized with myocardial infarction. JAMA. 2004 Oct 6;292(13):1563-72. doi: 10.1001/jama.292.13.1563. PMID 15467058
- [Background] Garcia M, Almuwaqqat Z, Moazzami K, Young A, Lima BB, Sullivan S, Kaseer B, Lewis TT, Hammadah M, Levantsevych O, Elon L, Bremner JD, Raggi P, Shah AJ, Quyyumi AA, Vaccarino V. Racial Disparities in Adverse Cardiovascular Outcomes After a Myocardial Infarction in Young or Middle-Aged Patients. J Am Heart Assoc. 2021 Sep 7;10(17):e020828. doi: 10.1161/JAHA.121.020828. Epub 2021 Aug 25. PMID 34431313
- [Background] Graham GN, Jones PG, Chan PS, Arnold SV, Krumholz HM, Spertus JA. Racial Disparities in Patient Characteristics and Survival After Acute Myocardial Infarction. JAMA Netw Open. 2018 Nov 2;1(7):e184240. doi: 10.1001/jamanetworkopen.2018.4240. PMID 30646346
- [Background] Bucholz EM, Ma S, Normand SL, Krumholz HM. Race, Socioeconomic Status, and Life Expectancy After Acute Myocardial Infarction. Circulation. 2015 Oct 6;132(14):1338-46. doi: 10.1161/CIRCULATIONAHA.115.017009. Epub 2015 Sep 14. PMID 26369354
- [Background] Udell JA, Desai NR, Li S, Thomas L, de Lemos JA, Wright-Slaughter P, Zhang W, Roe MT, Bhatt DL. Neighborhood Socioeconomic Disadvantage and Care After Myocardial Infarction in the National Cardiovascular Data Registry. Circ Cardiovasc Qual Outcomes. 2018 Jun;11(6):e004054. doi: 10.1161/CIRCOUTCOMES.117.004054. PMID 29848476
- [Background] Rao S, Jamal Siddiqi T, Khan MS, Michos ED, Navar AM, Wang TJ, Greene SJ, Prabhakaran D, Khera A, Pandey A. Association of polypill therapy with cardiovascular outcomes, mortality, and adherence: A systematic review and meta-analysis of randomized controlled trials. Prog Cardiovasc Dis. 2022 Jul-Aug;73:48-55. doi: 10.1016/j.pcad.2022.01.005. Epub 2022 Feb 1. PMID 35114251
- [Background] Yusuf S, Joseph P, Dans A, Gao P, Teo K, Xavier D, Lopez-Jaramillo P, Yusoff K, Santoso A, Gamra H, Talukder S, Christou C, Girish P, Yeates K, Xavier F, Dagenais G, Rocha C, McCready T, Tyrwhitt J, Bosch J, Pais P; International Polycap Study 3 Investigators. Polypill with or without Aspirin in Persons without Cardiovascular Disease. N Engl J Med. 2021 Jan 21;384(3):216-228. doi: 10.1056/NEJMoa2028220. Epub 2020 Nov 13. PMID 33186492
- [Background] Castellano JM, Sanz G, Penalvo JL, Bansilal S, Fernandez-Ortiz A, Alvarez L, Guzman L, Linares JC, Garcia F, D'Aniello F, Arnaiz JA, Varea S, Martinez F, Lorenzatti A, Imaz I, Sanchez-Gomez LM, Roncaglioni MC, Baviera M, Smith SC Jr, Taubert K, Pocock S, Brotons C, Farkouh ME, Fuster V. A polypill strategy to improve adherence: results from the FOCUS project. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2071-82. doi: 10.1016/j.jacc.2014.08.021. Epub 2014 Sep 1. PMID 25193393
- [Background] Wang TJ. The Polypill at 20 - What Have We Learned? N Engl J Med. 2022 Sep 15;387(11):1034-1036. doi: 10.1056/NEJMe2210020. Epub 2022 Aug 26. No abstract available. PMID 36018010
- [Background] Roshandel G, Khoshnia M, Poustchi H, Hemming K, Kamangar F, Gharavi A, Ostovaneh MR, Nateghi A, Majed M, Navabakhsh B, Merat S, Pourshams A, Nalini M, Malekzadeh F, Sadeghi M, Mohammadifard N, Sarrafzadegan N, Naemi-Tabiei M, Fazel A, Brennan P, Etemadi A, Boffetta P, Thomas N, Marshall T, Cheng KK, Malekzadeh R. Effectiveness of polypill for primary and secondary prevention of cardiovascular diseases (PolyIran): a pragmatic, cluster-randomised trial. Lancet. 2019 Aug 24;394(10199):672-683. doi: 10.1016/S0140-6736(19)31791-X. PMID 31448738